CLINICAL TRIAL: NCT04391231
Title: HEMolysis in a Percutaneous Axial Flow Left Ventricular Assist Device, Effects of Pentoxifylline in a Randomized Controlled Trial
Brief Title: HEMolysis in a Percutaneous Axial Flow LVAD, Effects of Pentoxifylline in a Randomized Controlled Trial
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Initially the study was underfunded; then, the device we planned to use was changed and the new pump significantly reduced hemolysis.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Dominic Emerson, MD, Staff Physician, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSMC - STUDY00000179
Record Dates: First submitted 2020-05-07; First posted 2020-05-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2022-09

CONDITIONS: Hemolysis Intravascular; Acute Decompensated Heart Failure
Keywords: CHF; Hemolysis; Impella
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Intervention Model Description: This study will be a double-blinded randomized placebo-controlled study to determine the efficacy of Pentoxifylline in reducing RBC hemolysis caused by Impella support.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be a double-blinded randomized placebo-controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentoxifylline Arm (Experimental): Pentoxifylline (in suspension with SyrSpend SF)
  Interventions: Drug: Pentoxifylline Oral Product
- Placebo Arm (Placebo Comparator): Placebo (SyrSpend SF only)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline Oral Product — Blinded Pentoxifylline (in suspension with SyrSpend SF)
  Arms: Pentoxifylline Arm
Drug: Placebo — Placebo (SyrSpend SF only)
  Arms: Placebo Arm

SUMMARY:
Temporary mechanical circulatory support devices are increasingly used for short-term support in patients with decompensated cardiogenic shock. Recently, a new axial flow pump has become widely available with the Impella System. The Impella has been FDA approved for short term usage. Hemolysis, however, has been a common complication that has increased morbidity and mortality in this patient population.

It is hypothesized that a major source of hemolysis in this patient population is shear stress experienced by red blood cells (RBC) as they travel through the pump device. In addition to causing RBC loss and potential anemia, the hemolysis has multiple other downstream consequences including creation of a pro-thrombotic environment leading to clot formation and potential device failure and secondary end organ dysfunction (renal and liver failure). Due to the significant effects of hemolysis in this population, a great deal of interest has been recently focused on addressing this problem, but as of yet no durable solutions exist.

Pentoxifylline improves red blood cell deformability and reduces blood viscosity. It is hypothesized here that administering Pentoxifylline to patients in CS who require temporary MCS will decrease the amount of shear stress related hemolysis through the improved deformability and durability of RBCs. We propose to perform a double-blinded randomized controlled trial in patients who undergo an axillary Impella 5.0 insertion for acute decompensated heart failure. There will be a control group who receives a placebo and the treatment group who receives pentoxifylline. Labs will be drawn to monitor hemolysis which is our current standard protocol for the life of the device to determine the efficacy of pentoxifylline in decreasing hemolysis in this patient population.

DETAILED DESCRIPTION:
Subjects will be screened prior to Impella device implant for eligibility. Informed consent will be obtained from eligible subjects. After implant of their Impella Device (5.0/5.5), results of laboratory tests (plasma free hemoglobin & lactate dehydrogenase levels) every 12 hrs for the first 3 days and then daily thereafter. Subjects will receive study medication every 6 hrs from device implant until device explant, death or Day 30 occurs. Impella therapy, concomitant medications and adverse events will be collected until the same. Subjects that don't qualify or opt out of participating will not receive the study medication. The data being collected for the study is based on routine standard of care. The difference between the SOC Impellas subjects and the study patients is the addition of Pentoxifylline being administered along with their SOC medications.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years of age
* Heart failure patients who undergo axillary Impella 5.0 or 5.5 insertion for acute decompensated heart failure

Exclusion Criteria:

* Concomitant temporary mechanical circulatory support (ECMO, RVAD)
* Heparin induced thrombocytopenia
* Recent cerebral and/or retinal hemorrhage or in patients who have
* Previous intolerance to Pentoxifylline or methylxanthines such as caffeine, theophylline, and theobromine
* Women who are currently pregnant, nursing or planning on becoming pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction in REBC hemolysis | Up to 30 Days post-device implant
  Measured by change in plasma free hemoglobin and lactate dehydrogenase levels

SECONDARY OUTCOMES:
hemolysis requiring adjustment of device speed settings | Up to 30 Days post-device implant
  Measured by change in plasma free hemoglobin and lactate dehydrogenase levels
device malfunction | Up to 30 Days post-device implant
  Impella system malfunction requiring intervention or device replacement
duration of Impella support | Up to 30 Days post-device implant
  Hours/days of Impella use
bleeding | Up to 30 Days post-device implant
  As assessed by drop in blood count
infection | Up to 30 Days post-device implant
  Assessed by fever and changes in laboratory assessments
death | Up to 30 Days post-device implant
  morbidity from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Domininc Emerson, MD, Principal Investigator — Cedars-Sinai Medical Center; Smidt Heart Institute
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lima B, Kale P, Gonzalez-Stawinski GV, Kuiper JJ, Carey S, Hall SA. Effectiveness and Safety of the Impella 5.0 as a Bridge to Cardiac Transplantation or Durable Left Ventricular Assist Device. Am J Cardiol. 2016 May 15;117(10):1622-1628. doi: 10.1016/j.amjcard.2016.02.038. Epub 2016 Mar 4. PMID 27061705
- [Background] Katz JN, Jensen BC, Chang PP, Myers SL, Pagani FD, Kirklin JK. A multicenter analysis of clinical hemolysis in patients supported with durable, long-term left ventricular assist device therapy. J Heart Lung Transplant. 2015 May;34(5):701-9. doi: 10.1016/j.healun.2014.10.002. Epub 2014 Nov 4. PMID 25582036
- [Background] Badiye AP, Hernandez GA, Novoa I, Chaparro SV. Incidence of Hemolysis in Patients with Cardiogenic Shock Treated with Impella Percutaneous Left Ventricular Assist Device. ASAIO J. 2016 Jan-Feb;62(1):11-4. doi: 10.1097/MAT.0000000000000290. PMID 26418208
- [Background] Ravichandran AK, Parker J, Novak E, Joseph SM, Schilling JD, Ewald GA, Silvestry S. Hemolysis in left ventricular assist device: a retrospective analysis of outcomes. J Heart Lung Transplant. 2014 Jan;33(1):44-50. doi: 10.1016/j.healun.2013.08.019. Epub 2013 Nov 14. PMID 24418733
- [Background] Nielsen VG, Pearson EC, Smith MC. Increased carbon monoxide production by hemeoxygenase-1 caused by device-mediated hemolysis: thrombotic phantom menace? Artif Organs. 2013 Nov;37(11):1008-14. doi: 10.1111/aor.12122. Epub 2013 Jul 19. PMID 23865494
- [Background] Jennings DL, Williams CT, Morgan JA. Pentoxifylline for the treatment of hemolytic anemia in a patient who developed recurrent gastrointestinal bleeding while on continuous-flow left ventricular assist device support. ASAIO J. 2013 Sep-Oct;59(5):526-7. doi: 10.1097/MAT.0b013e31829f0eb1. PMID 23896772
- [Background] Polonini HC, Silva SL, de Almeida TR, Brandao MAF, Ferreira AO. Compatibility of caffeine, carvedilol, clomipramine hydrochloride, folic acid, hydrochlorothiazide, loperamide hydrochloride, methotrexate, nadolol, naltrexone hydrochloride and pentoxifylline in SyrSpend SF PH4 oral suspensions. Eur J Hosp Pharm. 2016 Nov;23(6):352-358. doi: 10.1136/ejhpharm-2016-000903. Epub 2016 Mar 24. PMID 31156882
- [Background] Bansal A, Bhama JK, Patel R, Desai S, Mandras SA, Patel H, Collins T, Reilly JP, Ventura HO, Parrino PE. Using the Minimally Invasive Impella 5.0 via the Right Subclavian Artery Cutdown for Acute on Chronic Decompensated Heart Failure as a Bridge to Decision. Ochsner J. 2016 Fall;16(3):210-6. PMID 27660567